CLINICAL TRIAL: NCT04637568
Title: Comparative Evaluation of Paranasal Sinus Volumes Between Maxillary Deficiency Patients Requiring Le Fort Osteotomy and Control Patients
Brief Title: Paranasal Sinus Volumes of Maxillary Deficiency Patients Requiring Le Fort Osteotomy
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Poyzan Bozkurt, Associate Professor, Ankara University
Other Study IDs: AnkaraU 08/03
Record Dates: First submitted 2020-11-18; First posted 2020-11-19 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Maxillary Deficiency
Keywords: Maxillary Deficiency; Le Fort Osteotomy; Paranasal Sinus Volume; Computerized Tomography
MeSH Terms: conditions — Retrognathia | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Maxillary Deficiency: 59 CT scans of patients with maxillary deficiency requiring Le Fort osteotomy
  Interventions: Diagnostic Test: Computerized tomography
- Control: 61 CT scans of healthy patients
  Interventions: Diagnostic Test: Computerized tomography

INTERVENTIONS:
Diagnostic Test: Computerized tomography — Obtained CT scans involving the head region were analyzed retrospectively.

SUMMARY:
The present study aims to compare ethmoid, sphenoid and maxillary sinus volumes of patients with maxillary deficiency requiring Le Fort osteotomy with healthy patients, by employing computed tomography imaging. No accessible information could be found on this subject during literature search. The authors believe anatomical knowledge of these structures in patients with maxillary deficiency will influence all branches performing surgeries in these areas.

DETAILED DESCRIPTION:
The anatomy of the paranasal sinuses is important for many surgeon groups. The precise knowledge of such structures with variable anatomy will be important for the preservation of these structures and the management of complications in surgeries such as endoscopic sinus surgery and osteotomies involving the maxilla such as Le Fort osteotomies. The maxillomandibular complex is often affected by developmental problems and growth problems, and unilateral, bilateral, horizontal, vertical and / or transverse deficiencies are observed. Treatment of this complex is often performed by surgical intervention involving one or both jaws. In surgeries involving the maxilla, maxillary sinuses are affected by the surgery and affect the course of surgery. Paranasal sinuses are also very important structures for closely related endoscopic sinus surgeries. Detailed preoperative investigation is crucial for patient selection and hence desired outcome. Study was conducted in Ankara University Faculty of Dentistry with Ethical approval number:08/03. Computed tomography scans of 120 patients (59 maxillary deficiency patients and 61 healthy controls) were included in the study. CT scan indications for the group with maxillary deficiency was surgical preparation for Le Fort I osteotomy. The control group had no maxillary deficiency and CT images were obtained for several reasons such as temporomandibular disease, preparation for orthodontic treatment, obstructive sleep apnea and also paranasal sinus imaging Patients with a history of trauma in the midline skull base were excluded. Statistically significant results were obtained between groups for ethmoid and maxillary sinus volumes (left and right). Ethmoid and maxillary sinus volumes (left and right) were smaller in the Le Fort group. No statistically significant differences were present for sphenoid sinus volume of two groups and for the left and right maxillary sinus volumes in both groups.

ELIGIBILITY:
Inclusion Criteria for the study group:

- Maxillary deficiency (CT scans involving the head and paranasal sinuses, obtained for Le Fort I osteotomy).

Inclusion Criteria for the control group:

-Healthy patients. (CT scans involving the head and paranasal sinuses, obtained for several reasons such as temporomandibular disease, preparation for orthodontic treatment, obstructive sleep apnea and also paranasal sinus imaging, no maxillary deficiency).

Exclusion Criteria: Patients with a history of trauma in the midline skull base were excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population consisted of 58 male and 62 female participants, aged between 18-69.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Ethmoid sinus volumes | All measurements were taken twice by the same observers. The observers performed the study twice with an interval of 2 weeks to detect intra-observer variability.
  Ethmoid sinus volumes were calculated
Sphenoid sinus volumes | All measurements were taken twice by the same observers. The observers performed the study twice with an interval of 2 weeks to detect intra-observer variability.
  Sphenoid sinus volumes were calculated
Maxillary sinus volumes | All measurements were taken twice by the same observers. The observers performed the study twice with an interval of 2 weeks to detect intra-observer variability.
  Left and Right maxillary sinus volumes were calculated

CONTACTS AND LOCATIONS:
Overall Officials: Poyzan Bozkurt, Associate Professor, Principal Investigator — Ankara University
Locations (1):
- Ankara University Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No